CLINICAL TRIAL: NCT04931888
Title: Implementing and Evaluating a Wellness and Social-Emotional Learning Program for Refugee Children During the COVID-19 Pandemic: EMPOWER (Emotions Program Outside the Clinic and Wellness Education for Refugees)
Brief Title: Implementing and Evaluating a Social-Emotional Learning Program for Refugee Children During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Academic Pediatric Association (Industry); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000030455; KL2TR001862 (NIH)
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Social Emotional Wellness
Keywords: Refugee Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will receive the EMPOWER curriculum between the pre- and post-evaluations.
  Interventions: Behavioral: EMPOWER
- Waitlist (Other): The waitlist control arm will receive the EMPOWER curriculum after the evaluations. They will receive a second set of evaluations at the same time as the "post" evaluations of the control arm.
  Interventions: Behavioral: EMPOWER

INTERVENTIONS:
Behavioral: EMPOWER — EMPOWER is an adapted social emotional learning (SEL) and wellness education initiative delivered to a community of refugee families that was developed through a pre-pilot in the New Haven Afghan refugee community in 2020. Unlike traditional school-based SEL curricula, EMPOWER partners with community organizations to provide translated and trauma-informed wellness education to family units. The program combines in-person (socially distant) and remote delivery of culturally-informed physical, emotional, and medical wellness tools adapted from evidenced-based behavioral medicine, refugee trauma and recovery, and community health research.
  Other Names: Emotions Program Outside the Clinic and Wellness Education for Refugees

SUMMARY:
The overall goal of this overall goal is to pilot an adaptation of an established Social-Emotional Learning Program with novel wellness and COVID-19 safety components that are trauma-informed and culturally-specific in a resettled refugee community. In this pilot, "EMPOWER" (Emotions Program Outside the clinic and Wellness Education for Refugees), the study team will assess implementation outcomes (adoption, acceptability, and feasibility) of EMPOWER with refugee children and families during the COVID-19 pandemic through longitudinal evaluations and measurements of feasibility, acceptability, and attrition. The study team will also evaluate the impact of EMPOWER by assessing (a) children's social-emotional learning competence and (b) children's and family's COVID-19 knowledge.

DETAILED DESCRIPTION:
The major question that guides this research is: can an adaptation of an established Social-Emotional Learning (SEL) curriculum effectively improve Social-Emotional wellness for refugee children and their families? The hypothesis is that participation in this program will (a) improve children's SEL competence and (b) lessen stress and improve quality of life for refugee families.

The overall objective of this study is to establish and evaluate the preliminary efficacy and implementation of an adapted social-emotional learning (SEL) and Wellness Program for refugees: EMPOWER (Emotions Program Outside the clinic with Wellness Education for Refugees). To achieve the two aims of this study, the study team will conduct a wait-list controlled pilot to establish and evaluate the preliminary efficacy of participation in EMPOWER by assessing (a) children's SEL competence and (b) measures of mental health, stress, quality of life and wellness before and after participation in the program (Aim 1). Then, the study team will assess the implementation of EMPOWER with refugee children by using mixed methods to perform a summative evaluation of implementation outcomes-including fidelity, sustainability, and reach-in the Afghan refugee community (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* at least 1 year of schooling in the United States
* must speak: Pashto, Dari or English
* connected with the community organization: Elena's Light

Exclusion Criteria:

* inability to meet any of the requirements of the inclusion criteria

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Rosenberg, MD MHS, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosenberg J, McDonough Ryan P, Schaffer R, O'Brien C, Shabanova V, Ganjavi F, Sharifi M. Wait-List Controlled Pilot Trial of a Preventive Mental Health Intervention for Refugee Youth. J Immigr Minor Health. 2025 Oct;27(5):723-733. doi: 10.1007/s10903-025-01739-1. Epub 2025 Aug 9. PMID 40783623

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Family
Groups:
- Intervention - Child: The child respondents for the intervention group.
  The intervention arm received the EMPOWER curriculum between the pre- and post-evaluations.
  EMPOWER: EMPOWER is an adapted social emotional learning (SEL) and wellness education initiative delivered to a community of refugee families that was developed through a pre-pilot in the New Haven Afghan refugee community in 2020. Unlike traditional school-based SEL curricula, EMPOWER partners with community organizations to provide translated and trauma-informed wellness education to family units. The program combines in-person (socially distant) and remote delivery of culturally-informed physical, emotional, and medical wellness tools adapted from evidenced-based behavioral medicine, refugee trauma and recovery, and community health research.
- Intervention - Parent: The parent respondents for the intervention group.
  The intervention arm received the EMPOWER curriculum between the pre- and post-evaluations.
  EMPOWER: EMPOWER is an adapted social emotional learning (SEL) and wellness education initiative delivered to a community of refugee families that was developed through a pre-pilot in the New Haven Afghan refugee community in 2020. Unlike traditional school-based SEL curricula, EMPOWER partners with community organizations to provide translated and trauma-informed wellness education to family units. The program combines in-person (socially distant) and remote delivery of culturally-informed physical, emotional, and medical wellness tools adapted from evidenced-based behavioral medicine, refugee trauma and recovery, and community health research.
- Waitlist - Child: The child respondents for the waitlist group.
  The waitlist control arm received the EMPOWER curriculum and/or materials for EMPOWER after the evaluations. They will receive a second set of evaluations at the same time as the "post" evaluations of the control arm.
  EMPOWER: EMPOWER is an adapted social emotional learning (SEL) and wellness education initiative delivered to a community of refugee families that was developed through a pre-pilot in the New Haven Afghan refugee community in 2020. Unlike traditional school-based SEL curricula, EMPOWER partners with community organizations to provide translated and trauma-informed wellness education to family units. The program combines in-person (socially distant) and remote delivery of culturally-informed physical, emotional, and medical wellness tools adapted from evidenced-based behavioral medicine, refugee trauma and recovery, and community health research.
- Waitlist - Parent: The parent respondents for the waitlist group.
  The waitlist control arm received the EMPOWER curriculum and/or materials for EMPOWER after the evaluations. They will receive a second set of evaluations at the same time as the "post" evaluations of the control arm.
  EMPOWER: EMPOWER is an adapted social emotional learning (SEL) and wellness education initiative delivered to a community of refugee families that was developed through a pre-pilot in the New Haven Afghan refugee community in 2020. Unlike traditional school-based SEL curricula, EMPOWER partners with community organizations to provide translated and trauma-informed wellness education to family units. The program combines in-person (socially distant) and remote delivery of culturally-informed physical, emotional, and medical wellness tools adapted from evidenced-based behavioral medicine, refugee trauma and recovery, and community health research.
Period: Overall Study
Arm/Group | Intervention - Child | Intervention - Parent | Waitlist - Child | Waitlist - Parent
Started (Unit applied to children for consistency across columns. Although written as 0 units for parents to ensure the "total" column is correct, each parent is also from one family unit as well, corresponding to their child's family unit.) | 17; 5 Family | 5; 0 Family (The family unit is only applicable to the child arms of the study.) | 6; 3 Family | 3; 0 Family (The family unit is only applicable to the child arms of the study.)
Completed | 13; 3 Family | 3; 0 Family (The family unit is only applicable to the child arms of the study.) | 6; 3 Family | 3; 0 Family (The family unit is only applicable to the child arms of the study.)
Not Completed | 4; 2 Family | 2; 0 Family | 0; 0 Family | 0; 0 Family
Not completed — Excluded families participated in EMPOWER previously | 4 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants include parents and children (3 of intervention and 3 of waitlist control are parents). The intervention group included 3 families. The waitlist control group also included 3 families.
Groups:
- Intervention - Child: The Child respondents for the intervention group.
  The intervention arm will receive the EMPOWER curriculum between the pre- and post-evaluations.
  EMPOWER: EMPOWER is an adapted social emotional learning (SEL) and wellness education initiative delivered to a community of refugee families that was developed through a pre-pilot in the New Haven Afghan refugee community in 2020. Unlike traditional school-based SEL curricula, EMPOWER partners with community organizations to provide translated and trauma-informed wellness education to family units. The program combines in-person (socially distant) and remote delivery of culturally-informed physical, emotional, and medical wellness tools adapted from evidenced-based behavioral medicine, refugee trauma and recovery, and community health research.
- Intervention - Parent: The Parent respondents for the intervention group.
  The intervention arm will receive the EMPOWER curriculum between the pre- and post-evaluations.
  EMPOWER: EMPOWER is an adapted social emotional learning (SEL) and wellness education initiative delivered to a community of refugee families that was developed through a pre-pilot in the New Haven Afghan refugee community in 2020. Unlike traditional school-based SEL curricula, EMPOWER partners with community organizations to provide translated and trauma-informed wellness education to family units. The program combines in-person (socially distant) and remote delivery of culturally-informed physical, emotional, and medical wellness tools adapted from evidenced-based behavioral medicine, refugee trauma and recovery, and community health research.
- Waitlist - Child: The Child respondents for the intervention group.
  The waitlist control arm will receive the EMPOWER curriculum after the evaluations. They will receive a second set of evaluations at the same time as the "post" evaluations of the control arm.
  EMPOWER: EMPOWER is an adapted social emotional learning (SEL) and wellness education initiative delivered to a community of refugee families that was developed through a pre-pilot in the New Haven Afghan refugee community in 2020. Unlike traditional school-based SEL curricula, EMPOWER partners with community organizations to provide translated and trauma-informed wellness education to family units. The program combines in-person (socially distant) and remote delivery of culturally-informed physical, emotional, and medical wellness tools adapted from evidenced-based behavioral medicine, refugee trauma and recovery, and community health research.
- Waitlist - Parents: The Parent respondents for the intervention group.
  The waitlist control arm will receive the EMPOWER curriculum after the evaluations. They will receive a second set of evaluations at the same time as the "post" evaluations of the control arm.
  EMPOWER: EMPOWER is an adapted social emotional learning (SEL) and wellness education initiative delivered to a community of refugee families that was developed through a pre-pilot in the New Haven Afghan refugee community in 2020. Unlike traditional school-based SEL curricula, EMPOWER partners with community organizations to provide translated and trauma-informed wellness education to family units. The program combines in-person (socially distant) and remote delivery of culturally-informed physical, emotional, and medical wellness tools adapted from evidenced-based behavioral medicine, refugee trauma and recovery, and community health research.
- Total: Total of all reporting groups
Arm/Group | Intervention - Child | Intervention - Parent | Waitlist - Child | Waitlist - Parents | Total
Number analyzed (Participants) | 13 | 3 | 6 | 3 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.69 (0.76) | 37.67 (2.33) | 14.33 (3.51) | 7.50 (0.85) | 28.0 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 2 | 3 | 14
  Male | 6 | 1 | 4 | 0 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Afghan (Asian) | 13 | 3 | 6 | 3 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 3 | 6 | 3 | 25
Primary Language [Count of Participants; unit: Participants]
  Pashto | 9 | 1 | 5 | 2 | 17
  Dari | 4 | 2 | 1 | 1 | 8
Covid Knowledge Score [Mean (Standard Deviation); unit: units on a scale] — Number Correct out of 5 (yes/no) COVID-19 Knowledge Questions. Score range 0-5, with 0 being the lowest score (incorrect for all questions), and 5 being the highest score (correct for all questions. Population: Young children unable to answer questions were excluded
  units on a scale
    number analyzed (Participants) | 13 | 3 | 3 | 3 | 22
    (all) | 3.60 (0.22) | 4.33 (0.33) | 3.0 (1.0) | 3.33 (1.20) | 3.58 (0.26)
Trait Meta Mood Scale [Mean (Standard Deviation); unit: units on a scale] — Subscale from Trait Meta Mood Scale: Attention to Feelings Score, Maximum 35 (7 questions on a 1-5 Likert scale, with 35 being the highest score and 7 being the lowest score) Population: Participants who were parents were excluded, as responses reflected children's scores. Some responses were proxy responses (parent completed on behalf of child) and some were by children. If a parent expressed the child was too young to answer or have displayed answers to these questions, they did not complete the questions.
  units on a scale
    number analyzed (Participants) | 6 | 0 | 1 | 0 | 7
    (all) | 25.67 (1.43) |  | 25 (2) |  | 25.57 (1.23)
Pediatric Quality of Life Score [Mean (Standard Deviation); unit: units on a scale] — Scored subscales of: emotional, social, and school functioning. Ten total questions, each scored on a 0-4 Likert scale. Scores transformed to a 0-100 scale, with higher scores indicating a higher quality of life score. Population: Responses are only for child respondents, some with proxy respondents and some with child respondents.
  units on a scale
    number analyzed (Participants) | 13 | 0 | 5 | 0 | 18
    (all) | 70 (4.57) |  | 82.5 (4.87) |  | 73.47 (3.75)
Parent Afghan Symptom Checklist Score [Mean (Full Range); unit: units on a scale] — The Afhgan symptom checklist is a culturally-informed measure to evaluate distress and functioning in individuals from Afghanistan. We administered 21 of 22 questions to parents. Each question was scored on a scale of 1 to 5 (so minimum score (least distress) could be 21, and maximum score (most distressed) could be 105. Population: Only asked of parents. To save time and build trust, this exploratory measure was not asked on follow-up.
  units on a scale
    number analyzed (Participants) | 0 | 3 | 0 | 3 | 6
    (all) |  | 35.33 [25 to 56] |  | 43 [23 to 62] | 39.33 [23 to 62]

OUTCOME MEASURES:

1. Primary Outcome: Change in Social Emotional Competence
Description: Subscale from Trait Meta Mood Scale: Attention to Feelings Score, Maximum 35 (7 questions on a 1-5 Likert scale, with 35 being the highest score and 7 being the lowest score)
Time Frame: Baseline to 4 Weeks
Population: Children were excluded if they or their parents were unsure how to answer. The question was only asked of and/or about child participants (not parents)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Intervention - Child; Intervention Parent: The intervention arm received the EMPOWER curriculum between the pre- and post-evaluations.
  EMPOWER: EMPOWER is an adapted social emotional learning (SEL) and wellness education initiative delivered to a community of refugee families that was developed through a pre-pilot in the New Haven Afghan refugee community in 2020. Unlike traditional school-based SEL curricula, EMPOWER partners with community organizations to provide translated and trauma-informed wellness education to family units. The program combines in-person (socially distant) and remote delivery of culturally-informed physical, emotional, and medical wellness tools adapted from evidenced-based behavioral medicine, refugee trauma and recovery, and community health research.
- Waitlist - Child; Waitlist - Parent: The waitlist control arm received the EMPOWER curriculum and/or materials for EMPOWER after the evaluations. They will receive a second set of evaluations at the same time as the "post" evaluations of the control arm.
  EMPOWER: EMPOWER is an adapted social emotional learning (SEL) and wellness education initiative delivered to a community of refugee families that was developed through a pre-pilot in the New Haven Afghan refugee community in 2020. Unlike traditional school-based SEL curricula, EMPOWER partners with community organizations to provide translated and trauma-informed wellness education to family units. The program combines in-person (socially distant) and remote delivery of culturally-informed physical, emotional, and medical wellness tools adapted from evidenced-based behavioral medicine, refugee trauma and recovery, and community health research.
Arm/Group | Intervention - Child | Intervention Parent | Waitlist - Child | Waitlist - Parent
Number analyzed (Participants) | 12 | 0 | 2 | 0
units on a scale | 25.33 [20.83 to 29.83] |  | 20.00 [13.52 to 26.48] |

2. Primary Outcome: Change in COVID-19 Knowledge
Description: Number Correct out of 5 (yes/no) COVID-19 Knowledge Questions. Score range 0-5, with 0 being the lowest score (incorrect for all questions), and 5 being the highest score (correct for all questions).
Time Frame: Baseline to 4 Weeks
Population: Young children unable to answer questions were excluded
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Intervention - Parent: The intervention arm received the EMPOWER curriculum between the pre- and post-evaluations.
  EMPOWER: EMPOWER is an adapted social emotional learning (SEL) and wellness education initiative delivered to a community of refugee families that was developed through a pre-pilot in the New Haven Afghan refugee community in 2020. Unlike traditional school-based SEL curricula, EMPOWER partners with community organizations to provide translated and trauma-informed wellness education to family units. The program combines in-person (socially distant) and remote delivery of culturally-informed physical, emotional, and medical wellness tools adapted from evidenced-based behavioral medicine, refugee trauma and recovery, and community health research.
Arm/Group | Intervention - Child | Intervention - Parent | Waitlist - Child | Waitlist - Parent
Number analyzed (Participants) | 10 | 3 | 3 | 3
score on a scale | 4.50 [4.01 to 5.0] | 4.33 [3.48 to 5.19] | 4.00 [2.74 to 5.26] | 5 [5 to 5]

3. Secondary Outcome: Change in Quality of Life
Description: Scored subscales of: emotional, social, and school functioning. Ten total questions, each scored on a 0-4 Likert scale. Scores transformed to a 0-100 scale, with higher scores indicating a higher quality of life score.
Time Frame: Baseline to 4 Weeks
Population: Questions were only asked to or about children, not parents
Measure: Median (95% Confidence Interval); unit: score on a scale
Groups:
- Intervention - Child; Intervention - Parent: The intervention arm will receive the EMPOWER curriculum between the pre- and post-evaluations.
  EMPOWER: EMPOWER is an adapted social emotional learning (SEL) and wellness education initiative delivered to a community of refugee families that was developed through a pre-pilot in the New Haven Afghan refugee community in 2020. Unlike traditional school-based SEL curricula, EMPOWER partners with community organizations to provide translated and trauma-informed wellness education to family units. The program combines in-person (socially distant) and remote delivery of culturally-informed physical, emotional, and medical wellness tools adapted from evidenced-based behavioral medicine, refugee trauma and recovery, and community health research.
- Waitlist - Child; Waitlist - Parent: The waitlist control arm will receive the EMPOWER curriculum after the evaluations. They will receive a second set of evaluations at the same time as the "post" evaluations of the control arm.
  EMPOWER: EMPOWER is an adapted social emotional learning (SEL) and wellness education initiative delivered to a community of refugee families that was developed through a pre-pilot in the New Haven Afghan refugee community in 2020. Unlike traditional school-based SEL curricula, EMPOWER partners with community organizations to provide translated and trauma-informed wellness education to family units. The program combines in-person (socially distant) and remote delivery of culturally-informed physical, emotional, and medical wellness tools adapted from evidenced-based behavioral medicine, refugee trauma and recovery, and community health research.
Arm/Group | Intervention - Child | Intervention - Parent | Waitlist - Child | Waitlist - Parent
Number analyzed (Participants) | 13 | 0 | 5 | 0
score on a scale | 70 [60.35 to 79.65] |  | 82.5 [72.21 to 92.78] |

4. Secondary Outcome: Parent Afghan Symptom Checklist
Description: The Afhgan symptom checklist is a culturally-informed measure to evaluate distress and functioning in individuals from Afghanistan. We administered 21 of 22 questions to parents. Each question was scored on a scale of 1 to 5 (so minimum score (least distress) could be 21, and maximum score (most distressed) could be 105.
Time Frame: Only asked of parents. To save time and build trust, this exploratory measure was not asked on follow-up because of participant burden for questions.
Population: Only asked of parents. To save time and build trust, this exploratory measure was not asked on follow-up because of participant burden for questions.
Arm/Group | Intervention - Child | Intervention - Parent | Waitlist - Child | Waitlist - Parents
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Two months
Arm/Group | Intervention - Child | Intervention - Parent | Waitlist - Child | Waitlist - Parent
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/3 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/3 | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/13 | 0/3 | 0/6 | 0/3

LIMITATIONS AND CAVEATS:
Limitations included a smaller than expected sample size because of concurrent summer school opportunities. We also did not evaluate parental stress after participation because of this small sample size and question burden. Our translated instruments (Trait Meta Mood Scale, Peds-QL, COVID-19 questions) are early versions of translations, and will require formal validation in future studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT04931888/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT04931888/ICF_001.pdf